CLINICAL TRIAL: NCT05568563
Title: Comparison of Effectiveness of Pre-cooling With Ethyl Chloride Versus Honey in Alleviating Intra-oral Injection Pain in Adult Patients
Brief Title: Comparison of Effectiveness of Pre-cooling With Ethyl Chloride Versus Honey
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Altamash Institute of Dental Medicine (Other)
Responsible Party: Principal Investigator, Hira Abbasi, Principal Investigator, Altamash Institute of Dental Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ethyl Chloride versus Honey
Record Dates: First submitted 2022-10-02; First posted 2022-10-05 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Irreversible Pulpitis
MeSH Terms: interventions — Ethyl Chloride; Honey

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ethyl chloride (Experimental)
  Interventions: Drug: Ethyl chloride
- Honey (Experimental)
  Interventions: Other: Honey
- Control (No Intervention)

INTERVENTIONS:
Drug: Ethyl chloride — Ethyl chloride is an agent that is widely used in dental practice as the standard modality for pulp vitality tests .
  Arms: Ethyl chloride
Other: Honey — Honey is a natural dietary product
  Arms: Honey

SUMMARY:
Comparing Pre-cooling with Ethyl Chloride versus Honey in Alleviating Intra-oral injection pain in Adult patients

ELIGIBILITY:
Inclusion Criteria:

* No medical history
* Patients suffering from Symptomatic Irreversible Pulpitis requiring buccal infiltration

Exclusion Criteria:

* Patients having any medical conditions considered to affect patient safety or the quality of the study
* if they had any known hypersensitivity to local anaesthetics of amide type or any of the other contents in the substance used

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
To alleviate dental injection pain | immediately after completion of administration of oral local anesthetic infiltration within 60 seconds
  Post administration of oral local anesthetic infiltration pain will be measured by using Visual Analogue Scale(VAS) which is an 10-point scale from 0-10 where 0 represents no pain and 10 represents the worst pain measured

CONTACTS AND LOCATIONS:
Locations (1):
- Hira Danish, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No